CLINICAL TRIAL: NCT04451018
Title: Evaluation of Macro and Microcirculatory Arterial Condition of the Upper Limb in Insufficiently Renal Patients
Acronym: SYSTOE-HAIDI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.285; 2019-A02454-53 (Other: ID RCB)
Record Dates: First submitted 2020-02-14; First posted 2020-06-30 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Arteriopathy Upper Limb; Renal Insufficiency; Digital Pressure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: evaluation of arterial anomalies in upper limbs — evaluation of arterial anomalies in upper limbs with doppler ultrasound

SUMMARY:
Evaluation of macro and microcirculatory arterial condition of the upper limb in insufficiently renal patients

Hand ischemia affects 1.6 to 8% of patients with arteriovenous fistula (FAV) of hemodialysis in the upper limb. The diagnostic and therapeutic stakes are major as it concerns the functional prognosis of the hand and, to a lesser extent, vascular access for hemodialysis.

In some cases, the diagnosis of ischemic hemo-hijacking is evident, in other cases, the ischemic condition appears to be rather the result of uncompensated arteriatory of the upper limb or limbs. Echo-doppler exploration is usual for assessing vascular access but without validated formal criteria for arterial disease in the upper limbs, with fistula flow calculation and analysis of FAV hemodynamics. Compression manoeuvres on or under the FAV can also be performed. The pressures of the digital arteries are also indicated with non-consensual values found in the literature for the diagnosis of digital ischemia but with varying tools in terms of collection of measurements.

The main objective of this study is to collate the characteristics of arterial condition of the upper limbs of medium or severe renal patients, medium- or short-term candidates for kidney dialysis. The data collected will match the data of the arterial echodoppler as well as measures of pressures doppler laser and plethysmography. Candidates for dialysis tend to be older and polyvascular. A better assessment of the vascular condition of their upper limbs, including the diagnosis of advanced arterial disease, could eventually guide the choice of type of dialysis (compared to an indication of FAV).

DETAILED DESCRIPTION:
Prospective, monocentric study

The main objective of the research Description of the arterial condition of the upper limbs of kidney failure patients candidates for dialysis Primary Search Judgment Criterion: Description of the ultrasound characteristics of the arterial echo-doppler of the upper limbs.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal failure patient with nephrologist's decision to pre-dialysis Or Chronic renal insufficient patient with arteriovenous fistula of the upper limb and sign of digital ischemia (cold hand, digital ulcer, digital necrosis) Agreement on the study's non-opposition form Age above or equal 18 years Patient affiliated with a social security plan

Exclusion Criteria:

* Subject under guardianship or subject deprived of liberty Failure to obtain patient's consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic renal failure patient with nephrologist's decision to pre-dialysis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2025-06-17 (Estimated); Study Completion 2025-06-17 (Estimated)

PRIMARY OUTCOMES:
arterial condition of the upper limbs | 24 HOURS
  Description of the arterial condition with duplex ultrasound of the upper arteries: incompressibility or thrombosis of ulnar and/or radial arteries

CONTACTS AND LOCATIONS:
Overall Officials: Sophie BLAISE, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No